CLINICAL TRIAL: NCT00094367
Title: See Detailed Description
Brief Title: A Study Comparing Safety Of Abacavir And Lamivudine Administered Once-Daily As A Single Tablet Versus The Same Drugs Administered Twice-Daily As Separate Tablets (ALOHA Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101822
Record Dates: First submitted 2004-10-16; First posted 2004-10-18 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: HIV Infection
Keywords: 1592U89; GR109714; abacavir; lamivudine; fixed-dose combination; once-daily; twice-daily; HIV infection; naive
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine drug combination

INTERVENTIONS:
Drug: Abacavir/Lamivudine

SUMMARY:
This study was designed to evaluate if subjects who took 600 mg of abacavir and 300 mg of lamivudine once-daily as a single tablet were just as likely to have adverse events compared to subjects who took 300 mg of abacavir and 150 mg of lamivudine administered as separate tablets twice-daily.

DETAILED DESCRIPTION:
A phase IIIB randomized, open-label, multicenter, parallel-arm study to evaluate the short-term safety and tolerability of the abacavir/lamivudine fixed-dose combination tablet administered once-daily or the separate abacavir and lamivudine tablets administered twice-daily, as part of a three or four-drug regimen, in antiretroviral naive HIV-1 infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have HIV-1 infection.
* Had not received any prior HIV treatment for more than 14 days.
* At least 1000 copies of HIV-1 RNA.
* Willing to provide signed informed consent.

Exclusion Criteria:

* Enrolled in other investigational drug studies.
* Female subjects who are pregnant or breastfeeding.
* History of allergy or hypersensitivity to abacavir or lamivudine.
* Certain medical conditions that would make subjects ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2004-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The occurrence of treatment-limiting adverse events after starting study drugs.

SECONDARY OUTCOMES:
occurrence of abacavir HSR
completion of educational training
subject satisfaction with treatment
adherence to study medications
change in HIV-1 RNA from BL
change in CD4 measure from BL.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, PharmD, Study Director — GlaxoSmithKline
Locations (126):
- United States (126):
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Arleta, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Panorama City, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Salinas, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Glastonbury, Connecticut
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Stratford, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Inmokalee, Florida
  - GSK Investigational Site, Key West, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pampano, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Pompano Beach, Florida
  - GSK Investigational Site, Port Saint Lucie, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Riverdale, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Elgin, Illinois
  - GSK Investigational Site, Joliet, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Henderson, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Clinton, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Lowell, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Berkeley, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Saint Louis, Michigan
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, Englewood, New Jersey
  - GSK Investigational Site, Galloway, New Jersey
  - GSK Investigational Site, Hoboken, New Jersey
  - GSK Investigational Site, Jersey City, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Westfield, New Jersey
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Danville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin